CLINICAL TRIAL: NCT04214795
Title: The Effect of a Complete Course of Antenatal Steroids on Mortality and Morbidity of Preterm Infants
Brief Title: Antenatal Steroids Effect on Mortality and Respiratory Outcomes in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Manuel Sanchez Luna, Medical Doctor. Pediatric Profesor, Hospital General Universitario Gregorio Marañon
Other Study IDs: ANS- 2019
Record Dates: First submitted 2019-12-14; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Morbidity;Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants born after a complete course of antenatal steroids.: Preterm Infants born with less than 32 w GA whose mothers had received a complete course (two doses of celestone in the period between 24 hours and 7 days before delivery.
  Interventions: Other: Observational study. Postnatal variables are recorded
- Infants born without a complete course of antenatal steroids: Preterm Infants born with less than 32 w GA whose mothers did not received any dose of celestone or an uncompleted course (less than 24 hours or more than 7 days from delivery).
  Interventions: Other: Observational study. Postnatal variables are recorded

INTERVENTIONS:
Other: Observational study. Postnatal variables are recorded — Postnatal evolution is analyzed in both groups

SUMMARY:
The aim is to evaluate the impact of a complete course of antenatal steroids treatment on mortality and main morbidities in a current population of preterm infants.

DETAILED DESCRIPTION:
All infants admitted in the Neonatal Department born with less than 32 weeks of gestational age are included.

Data are prospectively recorded. Perinatal variables (Gestational age, materna condition at admission, antenatal steroids treatment, gender and results of histological analysis of the placenta) are recorded as well as respiratory status during hospitalization and morbidities at discharge. Results of neurodevelopment test performed at 24 months of corrected age are also included.

ELIGIBILITY:
Inclusion Criteria:

* All infants admitted in the NICU (with less than 6 hours after birth) born with less than 32+0 weeks of gestational age (GA).

Exclusion Criteria:

* Congenital malformations.
* premature infants in whom active resuscitation measures are not established.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants admitted with less than 6 hours after birth in the Gregorio Marañón Neonatal Department born with less than 32 weeks GA.
Sampling Method: Non-Probability Sample
Enrollment: 710 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | at hospital discharge, an average of 2-4 months.

SECONDARY OUTCOMES:
Number of participants with Bronchopulmonary dysplasia (BPD) diagnosis. | 36 weeks postmenstrual age
  BPD is considered as type 2 and 3 by consensus definition
Number of participants requiring Surfactant administration | in the first 3 days after birth
Number of participants that requires Mechanical ventilation. | during hospitalization, and average of 2-4 months
Number of participants with Neurodevelopment disability | performed at 24 months
  Scale of Psychomotor Development of Children (the Brunet-Lézine Scale). This scale consists of 150 items that are grouped around the following four areas: Posture (postural control or general motor skills), Coordination (psychomotor coordination), Language (comprehension and expression) and Sociability (social relations). The score of the items is binary (1/0) depending on whether the acquisition evaluated is achieved or not. The development age (ED) is obtained from the sum of the items. The result of dividing the age of development by postmenstrual age is the development quotient (CD). This calculation is practiced both for the set of items on the scale (global development quotient) and for each of the areas (partial development quotients).
  We have considered the value of the overall development quotient of less than 85 as the limit of normality, since it is a standard deviation below the expected development for its age.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Sánchez-Luna, MD, Study Director — Gregorio Marañón Hospital
Locations (1):
- Cristina Ramos-Navarro, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No